CLINICAL TRIAL: NCT02280642
Title: Alternate Dosing Schedules Study for HPV Vaccine
Brief Title: Alternate Dosing Schedules Study for HPV Vaccine (ADS)
Acronym: ADS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00014388_1; CDC#U36/CCU319276 CFDA 93.283
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Cervical Cancer; Genital Warts
Keywords: Human papillomavirus; Cervical cancer; Genital warts; Vaccine; Immunogenicity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Both doses on time: An on time dose 2 was defined as ≥ 30 days to ≤ 90 days after dose 1 and an on time dose 3 was defined as ≥ 60 days to ≤ 180 days after dose 2.
  Interventions: Biological: Both 2nd and 3rd doses on time
- Dose 2 delayed: A delayed dose 2 was defined as > 90 days after dose 1 and an on time dose 3 was defined as ≥ 60 days to ≤ 180 days after dose 2.
  Interventions: Biological: 2nd dose late and 3rd dose on time
- Dose 3 delayed: An on time dose 2 was defined as ≥ 30 days to ≤ 90 days after dose 1 and a delayed dose 3 was defined as >180 days after dose 2.
  Interventions: Biological: 2nd dose on time and 3rd dose late
- Both doses delayed: A delayed dose 2 was defined as > 90 days after dose 1 and a delayed dose 3 was defined as >180 days after dose 2.
  Interventions: Biological: Both doses late

INTERVENTIONS:
Biological: Both 2nd and 3rd doses on time
  Groups: Both doses on time
Biological: 2nd dose late and 3rd dose on time
  Groups: Dose 2 delayed
Biological: 2nd dose on time and 3rd dose late
  Groups: Dose 3 delayed
Biological: Both doses late
  Groups: Both doses delayed

SUMMARY:
The purpose of this study was to determine if delayed dosing of recombinant human papillomavirus (HPV) quadrivalent (Types 6, 11, 16, and 18) vaccine in 9-18 year old girls elicited an equivalent immune response (geometric mean titers to HPV 6,11,16, and 18 as measured one month after receipt of a 3rd dose of HPV vaccine) when compared to vaccine delivered according to the recommended dosing schedule.

This was a prospective observational study of healthy 9-18 year old female patients receiving either a second or third dose of HPV vaccine as part of their well child care. Immune responses to HPV types 6, 11, 16 and 18 were measured both before and 1 month after the third dose of HPV vaccine with the purpose of comparing the immune responses to HPV vaccine when administered at naturally occurring longer dosing intervals to the immune response to HPV vaccine when administered as routinely recommended.

In addition, girls receiving a 3rd dose of HPV vaccine as well as concomitantly administered vaccines by injection were randomized to receive either the HPV vaccine first or their concomitantly administered vaccines first. Pain following vaccination was assessed in each arm using the Faces Pain Scale - Revised.

Please note: This record refers only to the observational portion of the study. Please refer to NCT00862810 for the results of the randomized portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy, medically well female between the ages of 9 - 18 years. (Must be between 9 years and younger than 19 years of age) at time of enrollment
2. Must be receiving either a 3rd dose of HPV vaccine (All Groups) or a 2nd dose of HPV vaccine (Group 2 only)

   * For Group 1 - EITHER 1) The second dose of HPV vaccine must not have been administered and it must be within the specified dosing interval for the second dose of HPV vaccine (> 90 days since the first dose of HPV vaccine) OR 2) The second dose of HPV vaccine must have been administered > 90 days after the first dose of HPV vaccine and it must be within the specified dosing interval for the third dose of HPV vaccine (> 60 days - < 180 days since the second dose of HPV)
   * For Group 2 - The second dose of HPV vaccine must have been administered > 30 days and < 90 days after the first dose of HPV vaccine and it must be within the specified dosing interval for the third dose (> 180 days since the second dose of HPV)
   * For Group 3 - The second dose of HPV vaccine must have been administered > 30 days and < 90 days after the first dose of HPV vaccine and it must be within the specified dosing interval for the third dose (> 60 days - < 180 days since the second dose of HPV)
   * For Group 4- The second dose of HPV vaccine must have been administered > 90 days after the first dose of HPV of HPV vaccine and it must be within the specified dosing interval for the third dose (> 180 days since the second dose of HPV)
3. Ability and willingness to participate in the study by providing written informed assent. Verbal assent is acceptable for subjects less than 12 years of age.
4. Parent/guardian provides informed consent
5. Anticipated ability and willingness to complete all study visits and evaluations

Exclusion Criteria:

1. Unable to comply with the study protocol
2. Receipt of three or more doses of HPV vaccine or receipt of doses of HPV vaccine outside the pre-specified time windows
3. Receipt of blood and or blood products (including immunoglobulin) in the past 3 months or anticipated receipt during the study period
4. Receipt of a live virus vaccine (varicella virus containing vaccine, any measles, mumps, or rubella virus containing vaccine such as MMR, or yellow fever vaccine but not including live attenuated influenza virus vaccine) within 4 weeks of receipt of the 3rd dose of HPV vaccine or anticipated receipt of a live virus vaccine within 4 weeks after the 3rd dose of HPV vaccine
5. History of any physical, mental, or developmental disorder that study personnel believe may hinder a participant's ability to comply with the study requirements
6. History of malignancy or confirmed or suspected immunodeficient condition such as HIV infection
7. Receipt of or history of receipt of any medications or treatments that affect the immune system, such as immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity since six months prior to the first HPV vaccine dose. Receipt of long-term (greater than or equal to 2 weeks) potentially immunosuppressive corticosteroid use within six months prior to HPV vaccine dose 1 and enrollment or anticipated receipt during the study period. Specifically, potentially immunosuppressive corticosteroids are any parenteral corticosteroid, high dose (>800 mcg/day) beclomethasone dipropionate or equivalent medication. Nasal and topical steroids are allowed.
8. Current or former participation in HPV vaccine related research.
9. Receipt of an investigational or alternate HPV vaccine

Ages: 9 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent females attending primary care clinics in central North Carolina
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HPV 6 GMT | 1 month following 3rd dose of HPV vaccine
  Geometric mean titer (GMT) of antibody to HPV type 6
HPV 11 GMT | 1 month following 3rd dose of HPV vaccine
  Geometric mean titer (GMT) of antibody to HPV type 11
HPV 16 GMT | 1 month following 3rd dose of HPV vaccine
  Geometric mean titer (GMT) of antibody to HPV type 16
HPV 18 GMT | 1 month following 3rd dose of HPV vaccine
  Geometric mean titer (GMT) of antibody to HPV type 18

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Chapel Hill Pediatrics, Chapel Hill, North Carolina
  - Duke Children's Primary Care, Durham, North Carolina
  - Durham Pediatrics, Durham, North Carolina